CLINICAL TRIAL: NCT06518395
Title: The Degree of Knowledge and Attitude of Egyptian Nurses Regarding Emergency Management of Traumatic Dental Injuries: Cross-sectional Study
Brief Title: The Degree of Knowledge and Attitude of Egyptian Nurses Regarding Emergency Management of Traumatic Dental Injuries.
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hajar Adam, principle investigator, Cairo University
Other Study IDs: Egyptian nurses dental trauma
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Traumatic Dental Injuries
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire for The degree of knowledge and attitude. — Questionnaire for The degree of knowledge and attitude of Egyptian nurses regarding the emergency treatment of traumatic dental injuries

SUMMARY:
This study intends to evaluate medical and dental nurses' fundamental knowledge and attitude regarding the management of Traumatic Dental Injuries in Egypt.

DETAILED DESCRIPTION:
a master's degree student in the Department of Pediatric Dentistry ,Cairo University, will assess the degree of knowledge and attitudes of Egyptian Nurses regarding Emergency Management of Traumatic Dental Injuries for all the nurses who will be included in the study sample using soft and hard copies of questionnaire.

Data will be stored on the investigator's personal computer, secured with a password with backup for the data on Google Drive and hard copy.

The study results will be monitored regularly by the supervisors who will have full access to these interim results to make the final decision to terminate the study.

Auditing of the study design will be done by the evidence-based committee - Faculty of Dentistry - Cairo University.

Recruitment strategy will be through giving all medical and dental nurses at each hospital questionnaire forms to solve and return after explaining the items of the questionnaire to them.

The study size was calculated using StatCalc version 1.4.3 (Epi InfoTM, CDC, Atlanta, Georgia, USA) and it was a total of 371nurses.

Statistical analysis will be performed using Medcalc software, version 22 for windows (MedCalc Software Ltd, Ostend, Belgium).

ELIGIBILITY:
Inclusion Criteria:

* Egyptian Nurses who accepted to participate.

Exclusion Criteria:

* Egyptian Nurses who refused to participate.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical and dental Nurses in Egypt above 20 years of age.
Sampling Method: Probability Sample
Enrollment: 371 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
the degree of knowledge and attitude of Egyptian medical and dental Nurses about Emergency Management of Traumatic Dental Injuries. | 3 months
  the degree of knowledge and attitude of Egyptian medical and dental Nurses about Emergency Management of Traumatic Dental Injuries using Questionnaire as Measurement Method including Binary question (yes/no) and Multiple choice question.
  .

CONTACTS AND LOCATIONS:
Overall Officials: sherien B badr, professor, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
evaluate nurses' knowledge and attitude regarding management of TDIs in Egypt

REFERENCES:
- [Background] Caldas AF Jr, Burgos ME. A retrospective study of traumatic dental injuries in a Brazilian dental trauma clinic. Dent Traumatol. 2001 Dec;17(6):250-3. doi: 10.1034/j.1600-9657.2001.170602.x. PMID 11766091
- [Background] Andreasen JO, Andreasen FM, Skeie A, Hjorting-Hansen E, Schwartz O. Effect of treatment delay upon pulp and periodontal healing of traumatic dental injuries -- a review article. Dent Traumatol. 2002 Jun;18(3):116-28. doi: 10.1034/j.1600-9657.2002.00079.x. PMID 12110104
- [Background] Aldrigui JM, Abanto J, Carvalho TS, Mendes FM, Wanderley MT, Bonecker M, Raggio DP. Impact of traumatic dental injuries and malocclusions on quality of life of young children. Health Qual Life Outcomes. 2011 Sep 24;9:78. doi: 10.1186/1477-7525-9-78. PMID 21943368
- [Background] Andreasen JO, Andreasen FM, Andersson L, editors. Textbook and color atlas of traumatic injuries to the teeth. John Wiley & Sons; 2011 Dec 17.
- [Background] Andreasen JO, Andreasen FM, ed. Classifi cation, etiology and epidemiology. In: Textbook and color atlas of traumatic injuries to the teeth, 4th ed. Copenhagen: Blackwell Munksgaard; 2011. p. 218-19.
- [Background] Faus-Damia M, Alegre-Domingo T, Faus-Matoses I, Faus-Matoses V, Faus-Llacer VJ. Traumatic dental injuries among schoolchildren in Valencia, Spain. Med Oral Patol Oral Cir Bucal. 2011 Mar 1;16(2):e292-5. doi: 10.4317/medoral.16.e292. PMID 20711120
- [Background] Nourwali IM, Maddhar AK, Alsaati BH, Alhazmi RA, AlAyoubi SM, AlHarbi SS. Emergency management of dental trauma: a survey of public knowledge, awareness, and attitudes in Al-Madinah Al-Munawwarah. Clin Cosmet Investig Dent. 2019 Aug 27;11:279-284. doi: 10.2147/CCIDE.S205248. eCollection 2019. PMID 31695507
- [Background] Iyer SS, Panigrahi A, Sharma S. Knowledge and Awareness of First Aid of Avulsed Tooth among Physicians and Nurses of Hospital Emergency Department. J Pharm Bioallied Sci. 2017 Apr-Jun;9(2):94-98. doi: 10.4103/jpbs.JPBS_343_16. PMID 28717331